CLINICAL TRIAL: NCT03452215
Title: Impact of Mobile Application on Patient Knowledge of Pregnancy Topics
Brief Title: Mobile Application and Pregnant Patient Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Allison Reid, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01-18-30
Record Dates: First submitted 2018-01-30; First posted 2018-03-02 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy; Mobile Application
Keywords: Pregnancy; Mobile Phone Application

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental)
  Interventions: Behavioral: Mobile Phone Application Educational Resources; Behavioral: Mobile Phone Application GWG Tracker
- Control (Sham Comparator)
  Interventions: Behavioral: Mobile Phone Application Educational Resources

INTERVENTIONS:
Behavioral: Mobile Phone Application Educational Resources — Mobile Phone Application Educational Resources
Behavioral: Mobile Phone Application GWG Tracker — Mobile Phone Application GWG Tracker
  Arms: Study

SUMMARY:
Randomized controlled trial to investigate the impact of a pregnancy-specific mobile phone application on the knowledge of specific pregnancy topics and guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent (or 16-17 years of age with guardian present)
* Singleton gestation

Exclusion Criteria:

* Inadequate knowledge of English language
* Inability to read at or above 8th grade level
* Prior diagnosis of eating disorder

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy-specific topic/guideline questionnaire | Outcome assessed up to 23 weeks gestation
  Number of participants who correctly answer

SECONDARY OUTCOMES:
Pregnancy-specific questionnaire | Outcome assessed up to 23 weeks gestation
  Description of general patient population knowledge of pregnancy-specific topics and guidelines.
Gestational weight gain quantification | Outcome assessed through study completion, an average of 7 months
  Quantify total gestational weight gain with and without intervention from final documented weight during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No